CLINICAL TRIAL: NCT05381285
Title: Predictive Model of Mortality and Major Morbidity in Preterm Neonates in the Perinatal Period (Survival Model)
Brief Title: Survival Model for Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Cardiff University (Other); Swansea Bay University Health Board (Other)
Responsible Party: Sponsor
Other Study IDs: 20/AUG/7966; 287049 (Other: IRAS project ID); 22/PR/0147 (Other: REC reference)
Record Dates: First submitted 2022-04-01; First posted 2022-05-19 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Mortality; Morbidity;Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Non-interventional study

SUMMARY:
Study Title Predictive Model of Mortality and Major Morbidity in Preterm Neonates in the Perinatal Period Internal ref. no. / short title Survival Model Study Design Observational Population-based Cohort Study Planned Sample Size Retrospective analysis of Database Planned Study Duration 6-months Primary Objectives To derive a mathematical model for predicting mortality and the composite of mortality/major-morbidity before and immediately after birth in preterm infants Secondary Objectives Statistical Methodology and Analysis Mixed-model multivariable logistic regression analysis

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants born alive at or less than 34 weeks of gestation.
2. Born in Welsh maternity and admitted for care to a Welsh neonatal unit.
3. Mother normally resident in Wales

Exclusion Criteria

1. The mother is normally resident in England (detailed maternal data not available)
2. Congenital anomaly noted at birth (alters the natural probability of outcomes)
3. Duplicate episodes for an individual infant

Ages: 0 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The whole population of preterm infants born before 34 weeks of gestation for 8 years (2011-2018) in Wales will be included in the retrospective cohort.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 40-weeks
  In-hospital mortality
Mortality or major morbidity | 40-weeks
  In-hospital outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No